CLINICAL TRIAL: NCT02806037
Title: Utility of Intra-operative Image Guidance System for Missing Metastases
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: E15-166
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Metastatic to the Liver
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Intraoperatively, the surgeon will interrogate the liver with ultrasound. The time spent by the surgeon using the ultrasound is recorded. If all lesions seen on pre-op imaging were found, the patient does not have the Pathfinder Explorer system applied. If one or more lesions cannot be found, then the Pathfinder Explorer system is calibrated and a tracking device is attached to the ultrasound probe, which the surgeon will use to reattempt localization of the missing tumor. The Pathfinder Explorer system operates in real-time in conjunction with the ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* patient has one or more colorectal liver metastases, at least one of which is ≤1.5cm in maximal diameter on pre-operative cross sectional imaging
* undergoing liver resection and/or ablation

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the Hepatobiliary Clinic at Memorial Sloan-Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
localization rate of liver tumor | 1 year
  estimate the localization rate of Pathfinder to within +/-7%.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kingham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- [Derived] Kingham TP, Pak LM, Simpson AL, Leung U, Doussot A, D'Angelica MI, DeMatteo RP, Allen PJ, Jarnagin WR. 3D image guidance assisted identification of colorectal cancer liver metastases not seen on intraoperative ultrasound: results from a prospective trial. HPB (Oxford). 2018 Mar;20(3):260-267. doi: 10.1016/j.hpb.2017.08.035. Epub 2017 Sep 19. PMID 28935452
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/